CLINICAL TRIAL: NCT01345643
Title: A Randomized Controlled Clinical Trial of Transfusion Under the Guidance of West-China Perioperative Transfusion Score(WCPTS）for Massive Hemorrhagic Surgery
Brief Title: Clinical Trial of West-China Perioperative Transfusion Score (WCPTS）for Massive Hemorrhagic Surgery
Acronym: WCPTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ren Liao (Other)
Responsible Party: Sponsor-Investigator, Ren Liao, Associated Professor of Department of Anesthesiology, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCPTS110419
Record Dates: First submitted 2011-04-26; First posted 2011-05-02 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Transfusion Related Complications
Keywords: Transfusion; Hemoglobin level

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemoglobin level based on WCPTS (Experimental): According to WCPTS, the patient's hemoglobin level will be maintained not less than 7,8,9,or 10g/dL. Determination of whether a patient need red blood cells transfusion is based on WCPT Score.
  Interventions: Other: Transfusion trigger based on WCPTS
- Hemoglobin level 10g/dL (Active Comparator): The patient's hemoglobin level is maintained not less than 10g/dL perioperatively.
  Interventions: Other: Maintenance of hemoglobin level not less than 10g/dL

INTERVENTIONS:
Other: Maintenance of hemoglobin level not less than 10g/dL — The patient's hemoglobin level is maintained not less than 10g/dL perioperatively.
  Arms: Hemoglobin level 10g/dL
Other: Transfusion trigger based on WCPTS — Determination of whether a patient needs red blood cell transfusion or which hemoglobin level should be maintained is based on WCPTS
  Arms: Hemoglobin level based on WCPTS

SUMMARY:
Guidelines for blood transfusion have been issued for years. According to these guidelines, red blood cells (RBCs) transfusion should be given when the hemoglobin level is less than 6g/dL or 7g/dL and is unnecessary when the level is more than 10g/dL. However, in all the guidelines, the determination of whether RBCs should be administered when the hemoglobin level is in the range of 7~10g/dL is based on the judgment from anesthesiologists or surgeons. Index of transfusion trigger for patients with hemoglobin level between 7/dL and 10g/dL is necessary and important in clinical practice. Based on the aim of blood transfusion that maintain the balance of oxygen supply and oxygen consumption, the investigators hypothesize that index of transfusion trigger for patients with hemoglobin level between 7/dL and 10g/dL could be calculated by their history about heart and blood pressure, and routine monitoring parameters including pulse oximetry, temperature, and the use of vasoactive medications. To verify this hypothesis, the investigators present West China Perioperative Transfusion Score (WCPTS) for the trigger of transfusion according to the patient's history and monitoring parameters, and the investigators design a randomized controlled clinical trial to test this score.

DETAILED DESCRIPTION:
Surgery and trauma are the most common reasons for major blood loss, and blood transfusion provide guarantee for massive hemorrhagic surgery, especially orthopedic, cardiac, liver, and gynecologic procedures. On the other hand, blood transfusion is associated with many risks including hemolytic and nonhemolytic reactions, transfusion related acute lung injury, and others. Besides, blood is insufficient worldwide. How to eliminate allogeneic blood transfusion is an important part in clinical practice.

Guidelines for blood transfusion have been issued by many health institutions or organizations in different countries. According to these guidelines, red blood cells (RBCs) transfusion should be given when the hemoglobin level is less than 6g/dL or 7g/dL and is unnecessary when the level is more than 10g/dL. However, in all the guidelines, the determination of whether RBCs should be administered when the hemoglobin level is in the range of 7~10g/dL is based on the judgment from anesthesiologists or surgeons on the patient's condition including intravascular volume status, ongoing bleeding, any risk factors for vital organs ischemia or hypoxia, and so on. Index of transfusion trigger for patients with hemoglobin level between 7/dL and 10g/dL is necessary and important in clinical practice.

The aim of blood transfusion is to provide sufficient oxygen for the whole body, and to maintain the balance of oxygen supply and oxygen consumption. Factors associated with oxygen supply are hemoglobin level, cardiac output (CO), and oxygen saturation. Oxygen consumption is increased by the increase of metabolism, which could be reflected by increase of heart rate, blood pressure, and body temperature. If a patient's oxygen supply is decreased or oxygen consumption is increased, he will need a higher hemoglobin level to maintain the balance. Based on these findings, the investigators hypothesize that index of transfusion trigger for patients with hemoglobin level between 7/dL and 10g/dL could be calculated by their CO (reflected by the use of adrenalin), and routine monitoring parameters including pulse oximetry and core temperature.

West China Perioperative Transfusion Score (WCPTS)

The initial score is 7.

If a patient's cardiac output (CO) is normal without continuous infusion of adrenalin, or his SpO2 is more than 95%, or his core temperature is less than 38℃, he doesn't have any bonus point factor, and his score is 7.

If a patient's CO is maintained in normal range by continuous adrenalin infusion with concentration of less than 0.05μg/kg.min, or his SpO2 is 85~94%, or his core temperature is 38~40℃, his score should be added 1 point for every item mentioned above.

If a patient's CO is only maintained by continuous adrenalin infusion with concentration of more than 0.05μg/kg.min, or his SpO2 is less than 84%, or his core temperature is above 40℃, his score should be added 2 points for every item mentioned above.

For example, if a patient's CO is normal, his SpO2 is more than 95%, and his core temperature is 39℃,his WCPTS should be calcultaed as 7 plus 1 (core temperature is 39℃), and his final score is 8.

Here's another example, if a patient's CO is normal, his core temperature is less than 38℃, but he has COPD and his SpO2 is less than 84%, his score could be calculated as 7 plus 2(SpO2 is less than 84%), and his final score is 9.

Value of SaO2 is evaluated 5min after endotracheal intubation with inhalation of compressive air.

The initial score is 7，and the patient's score is calculated by 7 plus the sum of every item.

Score 7：To maintain the patient's Hb level not less than 7g/dL

Score 8：To maintain the patient's Hb level not less than 8g/dL

Score 9：To maintain the patient's Hb level not less than 9g/dL

Score 10 or >10：To maintain the patient's Hb level not less than 10g/dL

ELIGIBILITY:
Inclusion criteria

* Patients aged 15years to 70years.
* American Society of Anesthesiologists (ASA) physical status I, II, Ⅲ or Ⅳ.
* Undergoing elective spine surgery with estimated blood loss more than 800ml or 20% of the patient's whole blood volume.
* Glasgow Coma Scale (GCS) score of 15.
* Ability to communicate by telephone call.
* Informed consent has been signed by the patient or his legal guardian.

Exclusion criteria

* Declined to receive blood transfusion.
* Refuse to sign consent.
* Pregnancy.
* Psychopathy.
* Coagulopathy.
* Impairment of communication or cognition.
* Active participation in another trial where the primary endpoint follow-up is ongoing.
* Unwillingness or inability to comply with protocol procedures.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who received red blood cells transfusion | Up to 12 weeks.
  Proportion of patients who received red blood cells transfusion (Patients received red cells transfusion/ total number of the patients)
Transfusion volume of red blood cells | Up to 12 weeks.
  Volume of red blood cells transfused to the patients (units)

SECONDARY OUTCOMES:
All-cause mortality in 30 days post-operatively | Up to 30 days post-operatively.
  Death for any reason within 30 days post-operatively
In-hospital complications | Up to 12 weeks.
  In-hospital complications include: (1) Cardiac and pulmonary events such as cardiac arrest, arrhythmia, heart failure, pulmonary edema, etc. (2) Febrility without antibiotic treatment. (3) Infection needed antibiotic treatment. (4) Re-operation for bleeding. (5) Deep venous thrombosis. (6) Other complications.
Hb level at different time points | Up to 12 weeks.
  Hb level at admission, 1 day before surgery, during operation, 1,2,3 days after surgery, before discharge
Length of ICU stay and hospitalization | Up to 12 weeks.
  From admission to ICU to discharge from ICU
Costs of hospitalization and transfusion | Up to 12 weeks.
  All the medical costs.
Stitches removal time | Up to six months postoperatively
  The time period (days) from the day of operation to the day of stitches removal
Healing status of surgical incision | Up to six months postoperatively
  Healing status is divided into grade Ⅰ, Ⅱ, and Ⅲ. Grade Ⅰ was defined as the wound healing nicely without any adverse reaction, grade Ⅱ was defined as the inflammatory wound without the need of re-incision, and grade Ⅲ was defined as the wound suppurated with the need of re-incision for clearance.
Time to get recovery of daily life and/or working | Up to six months postoperatively
  Tthe time period (weeks) from the day of discharge to the day that patient get recovery of normal daily life and/or working during a six-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Study Director — Department of Anesthesiology, West China Hospital, Sichuan University; Jin Liu, M.D., Study Chair — Department of Anesthesiology, West China Hospital, Sichuan University
Locations (1):
- West China Hosptial, Sichuan University, Chengdu, Sichuan, China